CLINICAL TRIAL: NCT02801760
Title: Participation in a Biomedical HIV Prevention Clinical Trial: Perspectives of Younger and Older Young Men Who Have Sex With Men (YMSM) and Transgender Women Who Have Sex With Men
Brief Title: Self-Consent for PrEP Perspectives
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 137
Record Dates: First submitted 2016-03-23; First posted 2016-06-16 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-06

CONDITIONS: HIV; PrEP
Keywords: HIV; Self-Consent; PrEP; Autonomous Research Consent; Participation-associated Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects Currently or Previously Enrolled in ATN 110/ATN 113: Younger and older YMSM and transgender women who have sex with men, ages 15 through 22 years, inclusive, at the time of consent into the ATN 110 or ATN 113 study.
- Sub-Sample of Subjects to Complete Qualitative Interview: A sub-sample of subjects who completed the web-based survey and indicated willingness to complete the qualitative interview.

SUMMARY:
This study involves a one-time, web-based quantitative structured self-complete ("web-based") survey for all subjects and a qualitative semi-structured ("qualitative") interview for a selected sub-sample of subjects to evaluate the consent processes in association with research outcomes, specifically early adherence to Pre-exposure Prophylaxis (PrEP) and Human Immunodeficiency Virus (HIV) seroconversion at any point during participation in the ATN 110 or ATN 113 study.

DETAILED DESCRIPTION:
Decisional autonomy is a foundational, nearly inviolable principle of contemporary human subjects research. "Autonomy" refers to a deliberative outcome reflecting an individual's choice, outside of controlling influences of other agents. From the perspective of research participation decision-making, autonomy incorporates five elements of consent: competence; disclosure; understanding; voluntariness; and, consent. Adequate research consent processes are thought to be challenged by group-level qualities that define a "vulnerable population" in need of protection from coercion or undue influence. Age (typically less than age 18 in the United States) is a widely accepted status-defining vulnerability. Sexual minority identity or same-sex behavior does not define a "vulnerable" population but 45 Code of Federal Regulations (CFR) 46 subpart A (Common Rule) allows appropriate protections for other vulnerable populations as determined by an individual Institutional Review Board (IRB).

The specific aims of this study address issues within a larger domain of questions about the primacy of decisional autonomy, and associations of autonomous research consent and subsequent participation-associated outcomes. This mixed-methods study will enroll young men who have sex with men (YMSM) and transgender women who have sex with men who are currently or were previously enrolled in the ATN 110 or ATN 113 study.

Data from the web-based survey will be used to test hypotheses about the relationships between participant age, elements of the consent process, and two key participation outcomes (early adherence to PrEP, HIV seroconversion) in the ATN 110 or ATN 113 study. Data from the qualitative interview will be used to explore in further depth age-related vulnerability and disclosure vulnerabilities manifested for participants and whether/how they influenced ATN 110 and ATN 113 study outcomes. The interview will also assess decisional support and the benefits or harms associated with participation.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment into ATN 137, an individual must meet all of the criteria listed below.

* Is currently or was previously enrolled in the ATN 110 or ATN 113 study; and
* Is willing and able to provide informed consent via online informed consent form (ICF).

Exclusion Criteria:

To be considered eligible for enrollment, an individual must not meet any of the criteria listed below.

* Prematurely discontinued from the ATN 110 or ATN 113 study due to withdrawal of consent or inadvertent enrollment.
* Inability to complete the web-based quantitative structured self-completed survey in its entirety in a single sitting immediately after consent is provided.

Ages: 15 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: YMSM and transgender women who have sex with men who participated in the ATN 110 or ATN 113 study will be recruited to complete the one-time, web-based survey. Subjects who withdrew consent during their participation in the ATN 110 or ATN 113 study or were inadvertently enrolled will not be included in this study.
  A sub-sample of subjects who completed the web-based survey and indicated willingness to complete the qualitative interview will be selected to complete the qualitative interview. Selection will match subjects with high levels of PrEP adherence (> 4 doses/week) with those with low levels of PrEP adherence (< 4 doses/week). Attempt will be made to include all subjects that seroconverted.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Retrospective self-assessment of consent competence as assessed by completion of web-based survey | Day 1
Retrospective self-assessment of consent competence as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Retrospective self-assessment of consent disclosure as assessed by completion of web-based survey | Day 1
Retrospective self-assessment of consent disclosure as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Retrospective self-assessment of consent understanding as assessed by completion of web-based survey | Day 1
Retrospective self-assessment of consent understanding as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Retrospective self-assessment of consent voluntariness as assessed by completion of web-based survey | Day 1
Retrospective self-assessment of consent voluntariness as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Use of social support and information seeking in the consent process as assessed by completion of web-based survey | Day 1
Use of social support and information seeking in the consent process as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Experienced harms and benefits associated with autonomous research decision-making as assessed by completion of web-based survey | Day 1
Experienced harms and benefits associated with autonomous research decision-making as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Experiences with HIV testing and PrEP adherence technologies including home-based HIV testing Wisepill devices and text message adherence reminders as assessed by completion of web-based survey | Day 1
Experiences with HIV testing and PrEP adherence technologies including home-based HIV testing Wisepill devices and text message adherence reminders as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Post-ATN 110 or ATN 113 study PrEP use and experiences as assessed by completion of web-based survey | Day 1
Post-ATN 110 or ATN 113 study PrEP use and experiences as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent

SECONDARY OUTCOMES:
Types of vulnerabilities (i.e., age, sexual identity, sexual behavior, and race-related) that influenced ATN 110 and ATN 113 study outcomes as assessed by completion of web-based survey | Day 1
Types of vulnerabilities (i.e., age, sexual identity, sexual behavior, and race-related) that influenced ATN 110 and ATN 113 study outcomes as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Need for additional support in the decision making process for clinical trial participation as assessed by web-based survey | Day 1
Need for additional support in the decision making process for clinical trial participation as assessed by in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Self-assessment of adherence as assessed by web-based survey | Day 1
Self-assessment of adherence as assessed by in-depth interview with selected participants | One-time interview completed no more than 60 days after consent
Benefit or harm from participation as assessed by completion of web-based survey | Day 1
Benefit or harm from participation as assessed by completion of in-depth interview with selected participants | One-time interview completed no more than 60 days after consent

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, Ph.D., Study Chair — John Stroger Hospital of Cook County; J. Dennis Fortenberry, M.D., Study Chair — Indiana University School of Medicine
Locations (11):
- United States (11):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of Miami, Miami, Florida
  - University of Southern Florida College of Medicine, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Fenway Institute, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Childrens Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ATN Website — http://www.atnonline.org